CLINICAL TRIAL: NCT05284123
Title: The Impact of a Brief Self-Compassion Intervention on Shame and Mental Health Treatment-Seeking Among Distressed University Students
Brief Title: The Impact of a Self-Compassion Intervention on Shame and Mental Health Treatment-Seeking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Allison Kelly, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42483
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Psychological Distress
Keywords: Self-compassion; Mental health literacy; University students

STUDY DESIGN:
Intervention Model Description: 1/3 of the study participants (anticipated n=100) will be randomly assigned to the self-compassion intervention group, 1/3 of the participants (anticipated n=100) will be placed into the mental health literacy intervention group, and 1/3 of the study participants (anticipcated n=100) will be placed into the control group.
Who Masked: Participant
Masking Description: The participant will not know prior to their study participation that there are three different study conditions, and they will not find out which condition they were randomized to until the end of their study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-compassion intervention (Experimental): Brief (20-minute) workshop with a self-compassion writing exercise and information about mental health resources available to students.
  Interventions: Other: Self-compassion workshop
- Mental health literacy intervention (Experimental): Brief (20-minute) workshop with information and a written reflection about common mental disorders, and information about mental health resources available to students.
  Interventions: Other: Mental health literacy workshop
- Control (Active Comparator): Brief (7-minute) workshop with information about mental health resources available to students.
  Interventions: Other: Control workshop

INTERVENTIONS:
Other: Self-compassion workshop — The self-compassion workshop instructs participants to reflect on a source of shame, connect with their suffering related to it, and then direct feelings of support and understanding towards their suffering via a few brief writing tasks. This workshop also provides participants with basic information about mental health resources.
  Arms: Self-compassion intervention
Other: Mental health literacy workshop — The mental health literacy workshop provides participants with information about the symptoms and treatment of common mental disorders, and asks participants to reflect on what they learned through a couple brief writing tasks. This workshop also provides participants with basic information about mental health resources.
  Arms: Mental health literacy intervention
Other: Control workshop — The control workshop provides participants with basic information about mental health resources.
  Arms: Control

SUMMARY:
Untreated mental health problems can cause lasting harm to self-esteem, relationships, academics, productivity, and health. It is thus highly worrisome that only 18-36% of university students with significant mental health problems seek help. Many university campuses have responded to this mental health crisis by trying to increase students' mental health literacy (MHL), defined as "knowledge and beliefs about mental disorders which aid their recognition, management, or prevention''. Increasing MHL appears to increase knowledge about mental health services, but it does not increase actual treatment-seeking desire or action. One problem with this approach is that it falsely assumes that students struggling with their mental health will want to pursue services once they have learned more about mental disorders and the associated treatments available. However, most people with mental disorders do not initially recognize that they have a disorder and may dismiss information about mental disorders and mental health treatment as irrelevant. Feelings of shame are elevated in individuals with psychological disorders, and these feelings act as one of the strongest barriers to mental health treatment-seeking.Given the low rate of treatment-seeking on university campuses, research is needed to explore how best to facilitate mental health treatment seeking among distressed students, including those who may not self-identity as having a mental health problem. Research has yet to examine the potential role of self-compassion in relation to treatment-seeking behaviours. Self-compassion (SC) is conceptualized as responding to personal distress with gentleness and kindness in order to alleviate it, and it is negatively associated with shame. However, research has not yet explored whether the perceived benefits of SC in mitigating shame can affect mental health treatment-seeking outcomes. We propose that cultivating SC amongst psychologically distressed students will subsequently decrease shame, and thus, indirectly elevate willingness to seek mental health treatment. Thus, this study will examine the effects of a one-session SC workshop/intervention compared to a one-session MHL intervention on shame and mental health treatment-seeking. Participants will be distressed students recruited from the University of Waterloo, and will be randomly assigned to the SC intervention, MHL intervention, or control intervention.

DETAILED DESCRIPTION:
The study will consist of four online surveys. During the first survey (Part 1; baseline), participants will answer a set of questionnaires. During the second survey (Part 2; 1-4 days after Part 1), participants will first answer a set of questionnaires. Then, they will be randomized to a self-compassion intervention, a mental health literacy intervention, or a control intervention. Then, participants will answer more questionnaires immediately after completing the intervention. During the third survey (Part 3; 14-17 days after Part 2) and fourth survey (Part 4; 3 months-3 months+7 days after Part 2), participants will answer a set of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student at University of Waterloo with a SONA account
* Scored 8+ on Kessler Psychological Distress Scale (K6; screener scale)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
State Shame and Guilt Scale (shame subscale) | Change from pre-intervention to immediately post-intervention
  Self-report questionnaire with 5 questions on a 5-point Likert scale (scored 1-5). Total scores range from 5-25, with higher decrease in score indicative of less momentary shame.
Experience of Shame Scale | Change from baseline to 2 weeks and 3 months post-intervention
  Self-report questionnaire with 25 questions on a 4-point Likert scale (scored 1-4). Total scores range from 25-100, with higher decrease in score indicative of less shame.
Treatment-seeking intention questions (researcher-generated) | Change from baseline to immediately, 2 weeks, and 3 months post-intervention
  4 self-report questions to assess changes in intentions of seeking mental health treatment or resources.
Treatment-seeking behaviours questions (researcher-generated) | Change from baseline to immediately, 2 weeks, and 3 months post-intervention
  5 self-report questions to assess changes in mental health treatment-seeking behaviours.
Distress Disclosure Index | Change from baseline to immediately, 2 weeks, and 3 months post-intervention
  Self-report questionnaire with 12 questions on a 5-point Likert scale (scored 1-5). Total scores range from 12-60, with higher increase in score indicative of greater distress disclosure.

SECONDARY OUTCOMES:
Compassionate Engagement and Action Scale (adapted self-compassion subscale) | Immediately post-intervention
  Self-report questionnaire with 13 questions on a 10-point Likert scale (scored 1-10). Three questions are reverse-scored and not included in scoring. Total scores range from 10-100, with higher score indicative of greater momentary emotional engagement during intervention.
Kessler Psychological Distress Scale (K6) | Change from baseline to 2 weeks and 3 months post-intervention
  Self-report questionnaire with 6 questions on a 5-point Likert scale (scored 0-4). Total scores range from 0-24, with higher decrease in score indicative of less psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kelly, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No